CLINICAL TRIAL: NCT06920836
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Phase II Clinical Study to Evaluate the Efficacy and Safety of QR052107B Tablets in Patients With Subacute Cough
Brief Title: QR052107B Tablets in Patients With Subacute Cough of Phase Ⅱ Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QR052107B-YJXKS-2-1
Record Dates: First submitted 2025-03-28; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Cough
Keywords: Subacute Cough; selective P2X3 antagonist
MeSH Terms: conditions — Cough

STUDY DESIGN:
Intervention Model Description: Eligible subjects were randomized at a ratio of 1:1:1 into QR052107B 100 mg QD, QR052107B 400 mg QD and placebo groups and then entered the administration and observation period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatment assignment during the the administration and observation period will be kept blinded to participants, investigators, care providers, and outcome assessors if applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- QR052107B 100 mg QD (Active Comparator): Participants will be treated with one tablet of QR052107B 100mg, three tablets of placebo once daily for up to 9 days.
  Interventions: Drug: QR052107B 100 mg
- QR052107B 400 mg QD (Active Comparator): Participants will be treated with four tablets of QR052107B 100mg once daily for up to 9 days.
  Interventions: Drug: QR052107B 400 mg
- placebo QD (Placebo Comparator): Participants will be treated with four tablets of placebo once daily for up to 9 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QR052107B 100 mg — QR052107B 100 mg QD
  Arms: QR052107B 100 mg QD
Drug: QR052107B 400 mg — QR052107B 400 mg QD
  Arms: QR052107B 400 mg QD
Drug: Placebo — placebo QD
  Arms: placebo QD

SUMMARY:
The purpose of the study is to Evaluate the Efficacy and Safety of QR052107B 100mg， QR052107B 400mg in Patients with Subacute Cough.

DETAILED DESCRIPTION:
This study adopted a multicenter, randomized, parallel-group, double-blind and placebo-controlled design, and it was planned to enroll 270 patients with subacute cough following respiratory tract infection. After a screening period of 1-4 days, eligible subjects were randomized to the QR052107B 100 mg QD group, QR052107B 400 mg QD group and placebo group at a ratio of 1:1:1. The efficacy of QR052107B Tablets in the treatment of subacute cough was evaluated after 9 consecutive days of dosing. This study is divided into 3 stages: screening period, administration and observation period, and safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 (both inclusive), male or female.
2. Subjects with 18 kg/m2 ≤ BMI ≤ 30 kg/m2 at screening.
3. Subjects who have been diagnosed by the investigator with subacute cough (course of disease: 3-8 weeks) following respiratory tract infection.
4. Subjects who are willing to discontinue previous antitussives at screening.
5. Subjects who are willing to discontinue traditional Chinese medicines or Chinese patent medicines at screening.
6. Agreement to use at least one effective method of contraception during the study and for 3 months after the final dose.
7. Subjects who agree not to donate any sperm or egg during the study and for 3 months after the final dose.
8. Subjects who agree to sign the ICF and comply with all aspects of the study.

Exclusion Criteria:

1. Subjects with SPO2 ≤ 93% or significant polypnoea at rest during screening.
2. Subjects who have undergone chest X-ray or CT within 2 weeks before screening and have clinically significant lung lesions as judged by the investigator.
3. Subjects with cough and a large amount of thick phlegm that is difficult to expectorate and facing more safety risks in this study as judged by the investigator.
4. Subjects with acute respiratory tract infection (such as sputum purulent, pyrexia, white blood cell count increased or neutrophil count increased, and hs-CRP increased) as judged by the investigator at screening.
5. Subjects with infection in systems other than the respiratory system requiring systemic anti-infective therapy as judged by the investigator at screening.
6. Subjects with a history of chronic sinusitis, rhinitis allergic, seasonal cough and cough variant asthma (CVA), or with a history of systemic skin/mucosa allergy within 8 weeks before screening.
7. Subjects with a clear history of lung disorders (such as bronchial asthma, chronic obstructive pulmonary disease, pneumonia interstitial, pulmonary carcinoma and bronchiectasis) and unsuitable for this clinical study as judged by the investigator.
8. Subjects with severe or poorly controlled pre-existing diseases of various systems other than the respiratory system (such as liver disorders, chronic kidney disease, severe hematological diseases, chronic cardiac failure congestive [New York Heart Association (NYHA) Class III/IV], acute coronary syndrome, nervous system disorders including cerebrovascular and neuromuscular diseases, and metabolic diseases) and unsuitable for this clinical study as judged by the investigator.
9. Subjects with clinically significant abnormalities in clinical laboratory tests at screening and unsuitable for this clinical study as judged by the investigator, including but not limited to the following: alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT), serum total bilirubin (TBIL), and creatinine (Cr) > 200% × upper limit of normal (ULN).
10. History of alcohol or drug abuse in the past year.
11. Past or current history of major mental disorders.
12. Female subjects who are pregnant or lactating.
13. Subjects who are current smokers or have quit smoking within 6 months before screening.
14. Subjects who have participated in any other clinical trial within 3 months prior to screening, or are still in the safety washout period (< 5 half-lives) of the previous clinical trial on the first dosing day in this study, whichever is longer.
15. Presence of other factors that may increase the risk to subjects, affect the study results, or interfere with their participation in the whole study process, including but not limited to abnormal vital signs, physical examinations, ECGs and/or clinical laboratory tests, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
GMR of mean coughs per hour within 24 hours on D10 versus baseline | Baseline and day 10
  The geometric mean ratio (GMR) of mean coughs per hour within 24 hours on day10 versus baseline.

SECONDARY OUTCOMES:
GMR of mean coughs per hour within 24 h on D10 versus baseline in patients of ≥ 20 coughs per hour within 24 h at baseline | Baseline and day 10
  The geometric mean ratio of mean coughs per hour within 24 hours on day10 versus baseline in patients of ≥ 20 coughs per hour within 24 h at baseline.
GMR of mean coughs per hour within 24 h on D4 versus baseline in patients of ≥ 20 coughs per hour within 24 h at baseline | Baseline and day 4
  The geometric mean ratio of mean coughs per hour within 24 hours on day 4 versus baseline in patients of ≥ 20 coughs per hour within 24 h at baseline.
GMR of mean coughs per hour within 24 hours on D4 versus baseline | Baseline and day 4
  The geometric mean ratio of mean coughs per hour within 24 hours on day 4 versus baseline.
GMR of mean awake coughs per hour on D10 versus baseline | Baseline and day 10
  The geometric mean ratio of mean awake coughs per hour on day 10 versus baseline.
GMR of mean awake coughs per hour on D4 versus baseline | Baseline and day 4
  The geometric mean ratio of mean awake coughs per hour on day 4 versus baseline.
Change from baseline in cough severity VAS score on D4 and D10 | Baseline, day 4 and day10
  The changes in cough severity VAS score on D4 and D10 relative to baseline.
Change from baseline in LCQ-acute score on D4 and D10 | Baseline, day 4 and day10
  The changes in LCQ-acute score on D4 and D10 relative to baseline.
Change from baseline in sleep VAS score on D4 and D10 | Baseline, day 4 and day10
  The changes in sleep VAS score on D4 and D10 relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, MD, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No